CLINICAL TRIAL: NCT03076281
Title: A Phase II Study of Metformin, Doxycycline, or a Combination of Both Agents in Head and Neck Squamous Cell Carcinoma
Brief Title: Metformin Hydrochloride and Doxycycline in Treating Patients With Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient staff to conduct the trial
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16D.703; JT 9611 (Other: JeffTrial Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Larynx; LIP; Oral Cavity; Pharynx
MeSH Terms: conditions — Laryngeal Diseases | interventions — Metformin; Doxycycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride PO daily on days 1-3 and twice daily starting on day 4 to the day prior to surgery in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Metformin Hydrochloride
- Arm B (doxycycline) (Experimental): Patients receive doxycycline PO every 12 hours on days 1 to the day prior to surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxycycline
- Arm C (metformin hydrochloride, doxycycline) (Experimental): Patients receive metformin hydrochloride PO daily on days 1-3 and twice daily starting on day 4 to the day prior to surgery and doxycycline PO every 12 hours on days 1to the day prior to surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Metformin +Doxycycline

INTERVENTIONS:
Drug: Metformin Hydrochloride — Given orally
  Other Names: 1,1-Dimethylbiguanide Hydrochloride; 1115-70-4; 91485; Cidophage; Dimefor; Glucoformin; Glucophage; Glifage
  Arms: Arm A (metformin hydrochloride)
Drug: Doxycycline — Given orally
  Other Names: 17086-28-1; Doxycycline Monohydrate
  Arms: Arm B (doxycycline)
Drug: Metformin +Doxycycline — Given orally
  Arms: Arm C (metformin hydrochloride, doxycycline)

SUMMARY:
This randomized phase II trial studies how well metformin hydrochloride and doxycycline work in treating patients with head and neck squamous cell carcinoma that can be removed by surgery. Metformin hydrochloride may reduce the metabolic activity of cancer cells and of surrounding supportive tissue. Doxycycline may minimize toxic side effects of anti-cancer therapy. Giving metformin hydrochloride and doxycycline may work better in treating patients with head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if treatment with metformin hydrochloride (metformin), doxycycline, or a combination of metformin and doxycycline can increase the percentage of stromal cells that express CAV1 in patients with squamous cell carcinoma of the head and neck.

SECONDARY OBJECTIVES:

I. To determine the effect of metformin, doxycycline, or metformin and doxycycline treatment on the percentage of tumor cells that are apoptotic as determined by the TdT-Mediated dUTP Nick End Labeling Assay (TUNEL) assay, and express MCT4, MCT1, BGAL, and TOMM20 in squamous carcinoma of head and neck region tumor cells.

II. To assess safety and tolerability of metformin, doxycycline, or metformin and doxycycline treatment in subjects with squamous cell carcinoma of the head and neck.

TERTIARY OBJECTIVES:

I. To assess the effect of metformin, doxycycline, or metformin and doxycycline therapy on the metabolic profile of cancer cells and stroma using mass spectroscopy imaging (MSI) on paired samples, comparing metabolite profiles in the pre-treatment and post-treatment tumor samples.

II. To assess the effect of metformin, doxycycline, or metformin and doxycycline therapy on the metabolic state of the patient as characterized serologically by: erythrocyte sedimentation rate, exosome evaluation, metabolomics profile, and micro ribonucleic acid (RNA) expression profiles and physiologically by performing a nutritional assessment via a nutritionist-mediated 3-day dietary recall and comparing a patient's estimated dietary intake against their estimated caloric needs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of head and neck squamous cell carcinoma that is either biopsy proven or suspected based on history, physical, and or radiographic findings, and who are planned for definitive resection of the tumor without the use of neoadjuvant chemotherapy or radiation therapy at TJUH are eligible to participate.
2. Subjects must be ≥ 18 years of age at time of consent.
3. Patient must be able to swallow pills.
4. Patients with serum creatinine levels less than 1.5 mg/dL
5. Women of childbearing potential must have a negative urine or blood pregnancy test within 14 days of study enrollment.
6. Informed Consent: All subjects must be able to comprehend and sign a written informed consent document.
7. ECOG Performance status ≤1

Exclusion Criteria:

1. Subjects that do not have a baseline tumor specimen/biopsy prior to starting study medications.

   a. Tumor specimens do not need to be at Jefferson at time of eligibility determination. Tumor specimens held at outside institutions should be requested for analysis of pre-treatment tumor vs post-treatment tumor.
2. Subjects who are pregnant or breastfeeding, or may become pregnant during metformin and doxycycline administration.
3. Received prior cancer therapy for the HNSCC that is being resected.
4. Subjects on metformin or doxycycline for any reason during the preceding 4 weeks.
5. Diabetic subjects that are managed by taking metformin or insulin
6. Subjects who have received iodinated contrast dye must wait 12 hours prior to starting Metformin. If a CT scan with contrast is scheduled after screening and consent, the metformin cannot be taken until after the CT with contrast has been completed and they have waited 12 hours.
7. Patients with serum creatine ≥1.5 mg/dL
8. Patients with history of lactic or any other metabolic acidosis.
9. Patients with history of congestive heart failure stage III or greater.
10. Patients scheduled for definitive cancer surgical resection less than 7 days from beginning of study drug administration or greater than 6 weeks from beginning study drug administration.
11. Patients with history of hepatic dysfunction or hepatic disease and abnormal liver function tests defined as AST, ALT, Alk Phos, and or total bilirubin greater than 2.5 times the upper limit of normal. Patients who have a history of hepatic dysfunction or hepatic disease and normal liver function tests will be eligible to participate.
12. Patients with a current history (in the past 30 days) of heavy drinking which is defined in accordance with CDC definition as more than 8 drinks per week for women and more than 15 drinks per week for men. A standard drink contains .6 ounces of pure alcohol. Generally, this amount of pure alcohol is found in 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey). While on study, patients should limit their alcohol consumption to no more than 8 drinks per week for women and no more than 15 drinks per week for men.
13. Patient with prior allergic reaction to metformin, doxycycline, or any other tetracycline antibiotic in the past.
14. Patient is on medications that are contraindicated with metformin or doxycycline under current FDA recommendations. The following is a list of medications identified as class D (consider therapy modification) when treatment with metformin or doxycycline is considered:

    * Class D:

      * Bismuth Subsalicylate
      * Cimetidine
      * Iodinated cont

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Started | 3 | 2 | 2
Completed | 3 | 1 | 1
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline) | Total
Number analyzed (Participants) | 3 | 2 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 2
  >=65 years | 3 | 1 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of CFS Expressing Caveolin-1 at an Intensity of 1+ or Greater Assessed in Tumor-associated Stroma Cells by Immunohistochemistry
Description: Within-patient change in IHC scores will be analyzed using the Wilcoxon signed-rank test. Comparisons will be made between pretreatment and post-treatment within each of the cohorts. Caveolin-1 (CAV1) immunohistochemistry (IHC) will be performed on pre- and post-treatment tumor specimens. The mean percentage of fibroblasts expressing CAV1 will be compared before and after treatment.
Time Frame: Baseline to 30 days after last drug dose
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
percentage of cells | 32.5 [20 to 80] | 30 [30 to 60] | 32.5 [20 to 70]

2. Secondary Outcome: Incidence of Adverse Events as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Safety will be provided in descriptive tables as Incidence of adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 30 days after last drug dose: approximately1 year
Measure: Number; unit: adverse events
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
adverse events | 5 | 6 | 3

3. Secondary Outcome: Change in Percent of Tumor Cells Expressing MCT4, That Are TUNEL Positive and That Express BGAL
Description: Immunohistochemistry will be performed for Caveolin-1, TUNEL, BGAL, MCT1, MCT4, and TOMM20 on the pre- and post- treatment specimens and evaluated for staining distribution and intensity by two blinded pathologists.
Time Frame: Baseline to 30 days after last drug dose
Measure: Mean (Full Range); unit: Percentage of tumor cells
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
Percentage of tumor cells | 0 [0 to 0] | 12.5 [0 to 25] | 12.5 [0 to 25]

4. Secondary Outcome: Change in Percent of Tumor Cells Expressing MCT4, That Are TUNEL Positive and That Express MCT1
Description: as for outcome 3
Time Frame: Baseline to 30 days after last drug dose
Measure: Mean (Full Range); unit: Percentage of tumor cells
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
Percentage of tumor cells | 7.5 [0 to 15] | 7.5 [0 to 15] | 2.5 [0 to 5]

5. Secondary Outcome: Change in Percent of Tumor Cells Expressing MCT4, That Are TUNEL Positive and That Express MCT4
Description: as for outcome 3
Time Frame: Baseline to 30 days after last drug dose
Measure: Mean (Full Range); unit: Percentage of tumor cells
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
Percentage of tumor cells | 0 [0 to 0] | 12.5 [0 to 25] | 12.5 [0 to 25]

6. Secondary Outcome: Change in Percent of Tumor Cells Expressing MCT4, That Are TUNEL Positive and That Express TOMM20
Description: as for outcome 3
Time Frame: Baseline to 30 days after last drug dose
Measure: Mean (Full Range); unit: Percentage of tumor cells
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
Number analyzed (Participants) | 3 | 2 | 2
Percentage of tumor cells | 12.5 [0 to 25] | 12.5 [0 to 25] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm A (Metformin Hydrochloride) | Arm B (Doxycycline) | Arm C (Metformin Hydrochloride, Doxycycline)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Metformin Hydrochloride) (N=3) | Arm B (Doxycycline) (N=2) | Arm C (Metformin Hydrochloride, Doxycycline) (N=2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Metformin Hydrochloride) (N=3) | Arm B (Doxycycline) (N=2) | Arm C (Metformin Hydrochloride, Doxycycline) (N=2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Edema (General disorders) | 1 (1) | 1 (1) | 1 (2)
Neck Pain (General disorders) | 2 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to insufficient staff, which limited enrollment and overall data collection. While the outcome measures were completed for the few subjects enrolled, the small sample size and early termination prevent meaningful statistical interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03076281/Prot_SAP_000.pdf